CLINICAL TRIAL: NCT06542107
Title: Prediction of Weaning for Patients With Acute Brain Injury Undergoing Mechanical Ventilation
Brief Title: Weaning From Mechanical Ventilation in Patients With Acute Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Other Study IDs: WEAN ABI
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Ventilator Lung; Acute Brain Injury
Keywords: mechanical ventilation; acute brain injury; weaning
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute brain injury (ABI) patients frequently necessate intubation and invasive mechanical ventilation (IMV). While some ABI patients are capable of breathing spontaneously, which is one of the main criteria of extubation and weaning. However, the rate of extubation failure was significantly higher in ABI patients compared with non-neurological critical care patients. In patients who have failed one or several trials of extubation, tracheostomy is recommend according to the latest ESICM consensus. Tracheostomy can enhance comfort, improve pulmonary hygiene and decrease sedation requirement, which could facilitate the liberation from ventilator.

Numerous studies have explored the causes of weaning failure and provide various predictive models in guiding extubation and tracheostomy. Yet, due to limitations of such as small sample size or a lack of external validation, there is paucity of practical weaning algorithm tailored for ABI patients. The liberation from IMV in ABI patients still remains challenging with poor level of evidence in current guidelines or expert consensus.

We aim to describe the weaning outcomes in ABI patients, and further investigate the potential predictors of weaning success in ABI patients.

ELIGIBILITY:
Inclusion Criteria:

* acute brain injury
* age >=18 years
* invasive mechanical ventilation for at least 24 hours

Exclusion Criteria:

* tracheostomized before ICU admission
* pregnant or lactation
* with cervical spinal cord injury
* decision to receive palliative care within 24 hours of ICU admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU due to acute brain injury and treated with invasive mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 406 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
weaning success | up to 7-day period (ICU stay)
  successfully weaned from invasive ventilation according to WIND classification

SECONDARY OUTCOMES:
extubation | up to 7-day period (ICU stay)
  Extubation without the need for reintubation or death within a 7-day period, or upon ICU discharge, whichever occurs first

OTHER OUTCOMES:
tracheostomy | up to 7-day period (ICU stay)
  tracheostomy during ICU stay

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ling Liu, Nanjing, Jiangsu
  - Department of Critical Care Medicine, Zhongda Hospital, Nanjing